CLINICAL TRIAL: NCT06254807
Title: An Open-Label, Single-Arm Study of Autologous Anti-HER2 Chimeric Antigen Receptor Monocytes (CT-0525), in Participants With HER2 Over Expressing Solid Tumors
Brief Title: CAR-monocytes for the Treatment of HER2 Overexpressing Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Carisma Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Study 102
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-04

CONDITIONS: HER2-positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CT-0525 (Experimental): Cohort 1: 3 participants will be treated with a single IV administration of CT-0525 (3 billion CAR positive cells) on Day 1.
  Cohort 2: 3 participants will be treated with a single IV administration of CT-0525 (10 billion CAR positive cells) on Day 1.
  Interventions: Drug: CT-0525

INTERVENTIONS:
Drug: CT-0525 — Autologous monocyte engineered to contain an anti-HER2 chimeric antigen receptor

SUMMARY:
This is a first-in-human open-label study to evaluate the safety and tolerability, and manufacturing feasibility of anti-HER2 CAR-monocytes (CT-0525) in participants with locally advanced (unresectable) or metastatic solid tumors overexpressing HER2 whose disease has progressed on standard approved therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor tissue that is HER2-positive, following most recent therapy, by IHC using standard local assay resulting in 3+, or 2+ with confirmation by ISH testing. IHC and ISH assays and interpretation must follow the most recent ASCO/CAP guidelines and be performed in an accredited laboratory. Other tumor types (non-breast, non gastroesophageal) will be tested according to the breast cancer ASCO/CAP guidelines.
2. Histologically confirmed recurrent or metastatic solid HER2-positive tumor for which there are no available curative treatment options, AND after failure of the following systemic therapies used for the treatment of recurrent (unresectable) and/or metastatic disease:

   1. Any participant with HER2-positive breast or gastroesophageal cancers who has previously been treated with at least 2 FDA approved anti-HER2 therapies in the advanced/metastatic setting, including, but not limited to checkpoint inhibitors (i.e., PD-1/L1 inhibitors) and/or other targeted therapies for actionable molecular alterations (e.g., EGFR, ALK, ROS-1, BRAF, RET, MET, KRAS);
   2. Other HER2-positive tumor types must have progressed following treatment with at least 2 prior standard of care lines of therapy, including, but not limited to checkpoint inhibitors (i.e., PD-1/L1 inhibitors) and/or other targeted therapies for actionable molecular alterations (e.g., EGFR, ALK, ROS-1, BRAF, RET, MET, KRAS).
3. Participant must be willing and able to undergo on-study tumor tissue biopsy procedures to provide samples for biomarker analysis pre- and post-CT-0525 infusion:

   1. A participant whose tumor is not amenable to perform a safe post-baseline biopsy for the post-baseline translational studies may be allowed on the trial by mutual agreement of the Principal Investigator and Sponsor;
   2. Archived tumor tissue biopsy taken after progression on the most recent therapy is acceptable to be used in lieu of a pre-treatment biopsy for translational studies.
4. At least one measurable lesion (that will not be biopsied for eligibility and/or translational protocol requirements) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as assessed by the Investigator/site.
5. Eastern Cooperative Oncology Group (ECOG) Performance status 0-1 at screening.
6. Must have adequate hepatic function, as follows:

   1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels less than or equal to 3.0 x upper limit of normal (ULN) (less than or equal to 5 x ULN for participants with liver metastases) according to reference lab;
   2. Total bilirubin < 1.5 x ULN or direct bilirubin < 1.5 x ULN if total bilirubin is > 1.5 x ULN according to reference lab; for participants with Gilbert's syndrome total bilirubin < 3.0 mg/dL and direct bilirubin < 1.5 mg/dL.
7. Must have adequate cardiac function as follows:

   1. Class 0 or I/II cardiovascular disability according to the New York Heart Association Classification (Chavey, 2001);
   2. No history of unstable angina and/or myocardial infarction within 6 months prior to screening;
   3. Left ventricular ejection fraction (LVEF) less than or equal to 50% as determined by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA).
8. Must have an O2 saturation > 85%.
9. Pregnancy and Contraception/Barriers Female subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year, must be willing to use 1 highly effective method of birth control (as per Clinical Trial Facilitation Group [CTFG] guidance 2020), be surgically sterile, or abstain from heterosexual activity for the duration of the study through 120 days after the last dose of study medication. Refer to Appendix 4 for contraception guidance for female participants (Section 10.4).

   1. Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Refer to Appendix 4 for contraception guidance for female participants (Section 10.4).
   2. Male participants who are partnered with female participants of childbearing potential should be willing to use 1 highly effective method (as per Clinical Trial Facilitation Group [CTFG] guidance 2020) of birth control, be surgically sterile, or abstain from heterosexual activity for the duration of the study through 120 days after the last day of study medication.

Exclusion Criteria:

- Medical Conditions

1. Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study subjects of reproductive potential must have a negative urine pregnancy test at enrollment. The urine pregnancy test will need to be repeated prior to treatment if greater than 4 weeks has lapsed between the enrollment pregnancy test and treatment.
2. Known and previously documented human immunodeficiency virus (HIV) infection. Screening HIV test is not required in the absence of history or clinical suspicion.
3. Active hepatitis B or hepatitis C infection.
4. Diagnosis of immunodeficiency or exposure to systemic corticosteroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.

   1. Nasal or oral inhalers are permissible.
   2. Physiologic replacement doses of steroids (mineralocorticoid or less than or equal to a prednisone 10 mg daily dose) are permissible.
5. Any uncontrolled active medical disorder that would preclude participation as outlined.
6. Untreated or symptomatic central nervous system (CNS) metastases or cytology proven carcinomatous meningitis.
7. Participants with arrhythmias that are not stable on medical management, within 2 weeks of the Screening/Enrollment visit.
8. Known additional active and invasive malignancy within 5 years, other than the HER2 overexpressing malignancy being treated in this study.

   a. Exceptions include surgically cured non-melanoma skin cancers, noninvasive bladder tumors, or in situ breast or cervical cancer.
9. Uncontrolled acute bacterial, viral, or fungal infection (eg, blood culture positive less than or equal to 72 hours prior to study treatment) or any other clinically significant disease that, in the opinion of the investigator, would pose a risk to participant safety or interfere with the study evaluation, procedures or completion.

   Prior/Concomitant Therapy
10. Known history of allergy or hypersensitivity to human granulocyte colony-stimulating factors such as filgrastim or pegfilgrastim, or study product excipients including human serum albumin, Cryostor (DMSO or Dextran 40), or Plasma-Lyte.
11. Concurrent receipt of another anti-cancer therapy.

    Note: To be considered for inclusion in this study the following washout periods prior to apheresis must be completed as follows:
    1. Cytotoxic chemotherapy - 2 weeks;
    2. Tyrosine kinase/small molecule inhibitor - 2 weeks;
    3. Biologic therapy/monoclonal antibody - 4 weeks;
    4. Radiation therapy - 2 weeks;
    5. Prior investigational agent(s) - at least 5 half-lives of the agent in question, or 28 days, whichever is shorter prior to enrollment into the trial;
    6. With the exception of alopecia and the above Inclusion Criteria, participants must have recovered from prior treatment related toxicities with residual toxicity no greater than Grade 1 per CTCAE v.5.

    Prior/Concurrent Clinical Study Experience
12. Currently participating in or has participated in a study of an investigational agent or using an investigational device within 2 weeks of CT-0525 apheresis (4 weeks if investigational agent is a biologic/monoclonal antibody).

    1. Participants with previous cell therapy exposure may be eligible after discussion with the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Assess the safety and tolerability of CT-0525 by estimating the frequency and severity of adverse events in participants with HER2 overexpressing solid tumors. | Day 28
  Frequency and severity of adverse events including, but not limited to, estimating frequency and severity of Cytokine Release Syndrome (CRS).
Assess the feasibility of manufacturing CT-0525. | Baseline
  Percentage of products that pass release criteria among all manufactured products.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided